CLINICAL TRIAL: NCT00344240
Title: Aerobic Performance,Mobility Limitations and Exercise in Older Adults With Diabetes
Brief Title: Exercise and Activity Guidance in Older Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0966
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; exercise; activity guidance; health education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Health Education

INTERVENTIONS:
Behavioral: Functional circuit training with lifestyle behavior

SUMMARY:
The purpose of the project is to better understand how exercise and education will help mobility and health in older adults with diabetes. The investigators are trying to learn what type of exercises and classes are needed to help older adults stay active. This knowledge will eventually prove useful in helping patients and doctors understand what is needed to keep older adults with Type 2 diabetes as healthy as possible.

DETAILED DESCRIPTION:
1. Information and health screening: Interested persons are screened for eligibility and undergo a directed medical history and examination, echocardiogram (if not done within one year), limited ABI test, and maximal treadmill test with oxygen kinetics.
2. Measure fitness level at the beginning of the exercise training, at 10 and 20 weeks: DEXA scan, body fat analysis, strength and balance measurements, and blood tests.
3. Train for 10 weeks in a supervised small group format. Classes meet three times a week for an hour. Participants are randomly assigned to:

1) Flexibility and toning exercises + health education, or 2) Functional circuit training + home activities + tailored physical activity guidance.

4. Follow-up phone calls for an additional 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes on medications
* Age 60 or older
* Able to attend local class 3 times per week for 10 weeks

Exclusion Criteria:

* Ejection fraction <40%
* Symptomatic obstructive valvular disease (primarily aortic stenosis)
* Atrial fibrillation with poor rate control (particularly during exercise), or high grade AV block
* Substantial dementia (Folstein Mini Mental State Examination <24 out of 30)
* Blood tests suggesting severe renal (Cr>3.0) or hepatic (transaminases>4x normal) disease
* Alcohol intake >3 oz/day
* Hemiplegia or lower limb amputation
* Participating in regular exercise 2 or more hours per week.
* Significant orthopedic or musculoskeletal condition that limits weight bearing
* Acute medical conditions, such as acute flare-up of joint condition or infection
* Normal FBS in those with equivocal diabetes history (< 130)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Functional mobility performance
Physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Blaum, MD, Principal Investigator — University of Michigan. Ann Arbor Veterans Affairs Hospital
Locations (1):
- Mobility Research Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Lee PG, Ha J, Blaum CS, Gretebeck K, Alexander NB. Patterns of physical activity in sedentary older individuals with type 2 diabetes. Clin Diabetes Endocrinol. 2018 Apr 10;4:7. doi: 10.1186/s40842-018-0057-4. eCollection 2018. PMID 29662686
- See also: Mobility Research Center — http://www.med.umich.edu/geriatrics/moblab/index.htm